CLINICAL TRIAL: NCT01954537
Title: "Using Peak Core Temperature in Hot Preseason American Football Practice to Compare and Contrast Risk of Heat Illness at High School, College, and Professional Levels."
Brief Title: Comparing Risk of Heat Illness Based on Peak Core Temps During Preseason Football Camp Across 3 Different Age Levels
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1307M38681
Record Dates: First submitted 2013-09-18; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Exertional Heat Illness; Hydration Status
Keywords: Exertional heat illness; Hydration Status; Preseason football; heat stroke
MeSH Terms: conditions — Heat Stress Disorders; Heat Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Professional football players: Offensive and defensive professional football players ranging in age from 22 to 30 years old.
- Collegiate Football Players: Division III collegiate football players ranging in age from 20 to 23 years old.
- High School Football Players: High school football players ranging in age from 16 to 18 years old.

SUMMARY:
To collect field data in professional, collegiate, and high school football players to determine how they respond physiologically to the rigors of preseason training environment. Investigators will compare core temperature, hydration status, practice guidelines regarding rest and hydration, and baseline knowledge of heat illness and hydration among the three levels. The hypothesis is higher peak temperatures will be observed in the younger less experienced football players.

DETAILED DESCRIPTION:
Observations will occur over a 4-5 day period at the start of pre-season training camp. Researchers will meet with the high school volunteers and their parents to discuss the study and obtain informed consent prior to participating. Participants will swallow the HQInc CorTemp pill at least three hours (or late the night before) before practice. Temperature readings will be scanned every 15-30 minutes throughout practice. Pre and post practice weights will be recorded as well as urine specific gravity to help assess hydration status. Participants will also fill out a short 1 page questionnaire regarding their prior heat acclimatization, sleep habits, and baseline knowledge of hydration and heat illness. Protocol will be the same at all three age/competition levels.

ELIGIBILITY:
Inclusion Criteria:

* Football player on one of the teams from the pre-selected teams. Male.

Exclusion Criteria: based on being able to swallow HQInc CorTemp Pill

1. Any athlete weighing less than eighty (80) pounds.
2. Any athlete with any known or suspected diseases of the gastrointestinal tract.
3. Any athlete with impairment of the gag reflex.
4. Any athlete with previous gastrointestinal surgery.
5. Any athlete with history of problems with their esophagus.
6. Any athlete who might undergo an MRI scan before the temperature sensor has been eliminated from the body.
7. Any athlete with problems moving food through their gastrointestinal tract.
8. Any athlete having a cardiac pacemaker or other implanted electro medical device.

Min Age: 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be volunteers from the Minnesota Vikings Professional football team, Bethel University Division III football team, and Roseville High School football team.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Peak core body temperature | The first 3-4 days of preseason football practice for each cohort.
  Measured via HQInc ingestible core thermometer throughout practices.

SECONDARY OUTCOMES:
Hydration status before and after preseason football practice | Over first 3-4 days of each cohort's preseason camp.
  Measured via urine specific gravity and body weights before and after practice.
Baseline knowledge of hydration status and heat illness in football | Up to August 30th, 2013
  Athletes will be administered a 14 question survey covering various topics with regards to practice regulation, heat illness, and hydration.

CONTACTS AND LOCATIONS:
Overall Officials: Austin R Krohn, MD, Principal Investigator — University of Minnesota